CLINICAL TRIAL: NCT02793193
Title: Effect of Probiotics on Central Nervous System Functions in Humans
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University Hospital Tuebingen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PITN-GA-2013-607652
Record Dates: First submitted 2016-05-25; First posted 2016-06-08 (Estimated); Last update posted 2020-11-02 (Actual); Status verified 2016-05

CONDITIONS: Social Stress
MeSH Terms: interventions — Probiotics; Anti-Bacterial Agents

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Active (rifaximin/B.longum 1714) (Experimental)
  Interventions: Dietary Supplement: Probiotic; Drug: Antibiotic
- Placebo (Experimental)
  Interventions: Dietary Supplement: Placebo for antibiotic; Dietary Supplement: Placebo for probiotic

INTERVENTIONS:
Dietary Supplement: Probiotic — Probiotic B.longum 1714 will be donated by Alimentary Health Ltd. (Cork, Ireland) and each sachet contains 10 billion CFU
  Arms: Active (rifaximin/B.longum 1714)
Dietary Supplement: Placebo for antibiotic — The placebo supplementation is identical-looking to the antibiotic Xifaxan ®
  Arms: Placebo
Drug: Antibiotic — Antibiotic Xifaxan ® will be 200mg per tablet
  Arms: Active (rifaximin/B.longum 1714)
Dietary Supplement: Placebo for probiotic — The placebo identical-looking to the probiotic B.longum 1714
  Arms: Placebo

SUMMARY:
The gut-brain axis is described as being important in both, gut functions and central nervous system (CNS) functions. The microbiota in the gut plays an important role in this axis through neural, immune and endocrine systems. Previous studies have found altered gut microbiota (GM) composition could change the CNS functions in animals and humans. Probiotics were shown having positive effect on improving stress response in animals and stress related psychiatry in humans. The current study will investigate if probiotics can improve response to social stress in healthy participants and patients with irritable bowel syndrome (IBS), which is a stress-related disease, and whether this probiotic action can be counteracted by the locally acting antibiotic, Rifaximin. The investigators will use the Cyberball paradigram to induce social stress and magnetoencephalography (MEG) to record neural responses related to the social stress. The administration of the probiotics will be a new strategy for both the mental health management and treatment of gastrointestinal (GI) disorders in the future.

DETAILED DESCRIPTION:
Understanding the neural mechanisms underlying the experience of social stress may help to prevent the development of IBS and to help people to maintain their mental health. Social distress has been examined with the Cyberball paradigm in developing peers and children with autism spectrum disorders, people with social anxiety disorder and with borderline personality disorder. These studies provided researchers the clinical evidence and validity of the paradigm in patients . Here the investigators will examine the neural response of healthy volunteers to acute stress induced by the Cyberball game and if acute intervention with probiotics for 4 weeks can alleviate the stress response. The study will be firstly conducted on healthy volunteers whose GM will be disturbed by an antibiotic Rifaximin as to simulate IBS patients, to see their neural response to the social exclusion (Study 1). The second study will be conducted as a clinical trial in healthy volunteers to investigate the effect of the probiotic Bifidobacterium longum 1714 (Study 2).

Study 1 & 2 will be a randomized, double blind, double dummy design, during which the participants will visit the laboratory for 2 times (M1, M2,): measurement at baseline and after intervention. Intervention period lasts for 1 week in study 1 and 4 weeks in study 2.

In study 1, Group 1 will take Rifaximin for 1 week Group 2 will take Placebo for 1 week

In study 2, Group 1 will take B.longum 1714 for 4 weeks Group 2 will take Placebo for for 4 weeks

Participants will be not allowed to eat certain kinds of food. As mentioned in the exclusion criteria, participants will not eat probiotic/prebiotic containing food supplements, or potentially immune-enhancing dietary supplements either. The food to be avoided will be summarized on a list of probiotic/prebiotic containing food. Also, participants will be asked to record the food they take on each day during the intervention, by taking photos. Nutritional information about the food taken by the participants will be analyzed by using an online tool http://nutritiondata.self.com/.

Before the intervention period, each participant will need to complete questionnaires including a demographic questionnaire, the Patient Health Questionnaire (PHQ) and the Hospital Anxiety and Depression Scale (HADS). The PHQ is for excluding those healthy participants who suffer from psychiatry disorder(s) and for further analysis. The HADS, which will also be completed after each intervention period, aims to study the effect of the probiotic on anxiety and depression level in healthy participants and especially in IBS patients. Also, participants will receive a daily online questionnaire via email, including the Positive Affect and Negative Affect Scales, and questions about their level of stress, consumption of the study capsules, hours of sleep, IBS symptom and quality of life (QoL) (the last two are only for patients), etc. Through questionnaires, the investigators will record menstruation information of female participants for controlling confounders. Also, gender and age between healthy and patient groups will be matched as much as possible, since these factors could have an effect on the GM composition and the CNS functions.

Stool samples will be collected on the day participants come to a lab visit for measurements. The stool sample should be as fresh as possible, ideally collected in the morning of the visiting day. Fresh samples will be stored in RNA synthesis stabilization buffer at the time of collection. A centrifuged fecal pellet will be stored at -80°.

During the Magnetoencephalography measuring, before the Cyberball game, there will be a resting state session for 5 minutes. In this session participants will be studied in supine position. Participants will be instructed to move as little as possible and remain awake, while keeping their eyes closed. After the resting state recording the Cyberball game will start. The task of the game will be projected on a screen and participants will be asked to fixate the screen and hold a response box to get ready for the task. Magnetic fields will be measured with a 275-channel whole head magnetometer at a sampling rate of 1200 Hz. In order to overlay the brain activity derived from MEG on anatomical scans, a high-resolution (1 mm, isotropic) T1-weighted structural MR image will be acquired with an MPRAGE sequence with a 3-T MR scanner (University Hospital Tübingen, Tübingen, Germany).

7 participants will be needed in each experimental group in study 1, resulting in at least 14 in study 1. 20 participants will be needed in each experimental group in study 2, resulting in at least 40 in study 2. The recruitment of participants will be organized by the MEG center under the responsibility of Prof. Dr. Christoph Braun. The study will be announced on black boards in the Tübingen University Clinic and the campus of the University. Further announcements will be done via the University mailing list and the local newspaper. Each participant will be provided with detailed information about the aims of the investigation, the tasks and measurements. Participants will be informed about the possibility to cancel the examination at any time without cause or prejudice for her person. Investigation will be carried out only when written consent from the participants is obtained.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female volunteers aged 18 to 50 years.
2. Signed informed consent. Written informed consent will need to be obtained from all participants, and the protocol will be submitted to the Ethics Board of the Medical School for approval,
3. Participant is willing to comply with the study restrictions.
4. Participant has been a non-smoker for at least 3 months.
5. Participants with body mass index 18-30.

Exclusion Criteria:

1. Participants are current smokers,
2. Participants have chronic allergies,
3. Participants are unwilling to discontinue the consumption of probiotic- and prebiotic-containing foods or potentially immune-enhancing dietary supplements (i.e. prebiotics, probiotics, Echinacea, fish oil and vitamin E (>400 % of the RDA or .60 mg/d)),
4. Participants received an immune-suppressing intervention or have an immunosuppressive illness within the last year,
5. Participants have a psychiatric disorder (eg. depression, anxiety, dysthymia, panic disorder, disorder of mania or bipolar disorder, phobia, post-traumatic stress disorder, substance abuse, eating disorder) (only for recruiting healthy volunteers).
6. Participants received antibiotic therapy within the last 2 months of their study start date.
7. Participants have non-removable metal parts in the body such as: pacemaker, artificial heart valves, metal prostheses, implanted magnetic metal parts (screws), spiral, metal fragments / shrapnel, fixed braces, acupuncture needle, insulin pump, tattoos, eye shadow. Also, people with agoraphobia will be excluded.
8. Patients who do not meet the diagnosis criteria of IBS based on Rome I, II, or III (only for recruiting patients).

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 54 (Actual)
Dates: Start 2016-07; Primary Completion 2018-01 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
Neural response to social stress measured by Magnetoencephalography | 8 weeks

SECONDARY OUTCOMES:
Bacterial population levels in faecal samples | 8 weeks
Cortisol levels in blood samples | 8 weeks
Tryptophan levels in blood samples | 8 weeks
Score of the Hospital Anxiety and Depression Scale (HADS) | 8 weeks
  the RAND 36-Item Healthy Survey
Scores of the Positive and Negative Affect Scales (PANAS) | 8 weeks
Scores of the RAND 36-Item Healthy Survey | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Paul Enck, Prof. Dr., Principal Investigator — Department of Internal Medicine VI: Psychosomatic Medicine and Psychotherapy, University of Tuebingen
Locations (1):
- University Hospital Tuebingen MEG Center, Tübingen, Germany

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Wang H, Braun C, Enck P. Effects of Rifaximin on Central Responses to Social Stress-a Pilot Experiment. Neurotherapeutics. 2018 Jul;15(3):807-818. doi: 10.1007/s13311-018-0627-2. PMID 29713909